CLINICAL TRIAL: NCT00636974
Title: Minimum Local Anaesthetic Dose for Intrathecal Anaesthesia: a Randomised Comparison Between Levobupivacaine, Ropivacaine and Bupivacaine
Brief Title: A Randomised Comparison on the Dose Requirement Between, Levobupivacaine, Ropivacaine and Bupivacaine in Intrathecal Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KW/FR/05-025; HARECCTR0500056
Record Dates: First submitted 2007-12-19; First posted 2008-03-17 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Anesthesia, Conduction; Surgery
Keywords: Patients who are going to have regional anaesthesia for lower limbs surgery.; Leg Surgery.

INTERVENTIONS:
Procedure: Combined spinal epidural anaesthesia

SUMMARY:
To determine and compare the effective intrathecal dose of levobupivacaine, ropivacaine and bupivacaine for 50% of patients in lower limb surgery

ELIGIBILITY:
Inclusion Criteria:

* body weight=40-90kg,
* height higher than 145cm

Exclusion Criteria:

* Known hypersensitivity to amide local anaesthetics,
* patients who do not understand English and Chinese,
* Body mass index higher than 35 kg per sq metre

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2006-01; Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Sensory block at 12th thoracic dermatome or above and successful conduct of the lower limb surgery up to 50 minutes after the intrathecal injection of the study drug | 50 minutes after the intrathecal injection of the study drug

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yin Lee, Dr, Principal Investigator — Department of Anaesthesiology, Kwong Wah Hospital
Locations (1):
- Kwong Wah Hospital, Hong Kong, China